CLINICAL TRIAL: NCT03904069
Title: A Phase 1 Study Evaluating the Safety, Tolerability, and Efficacy of FLT3 Chimeric Antigen Receptor T-cell (CAR-T) AMG 553 in Subjects With FLT3-positive Relapsed/Refractory Acute Myeloid Leukemia.
Brief Title: Study Evaluating the Safety, Tolerability, and Efficacy of FLT3 CAR-T AMG 553 in FLT3-positive Relapsed/Refractory AML
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Following a recent cellular therapy strategy assessment, Amgen has decided to cancel study 20180091.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180091
Record Dates: First submitted 2019-03-21; First posted 2019-04-04 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
Keywords: Relapsed/refractory acute myeloid leukemia; Acute myeloid leukemia; Oncology/hematology; CAR T cell therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Comparison of different cell doses of AMG 553 (Experimental): Subjects will receive IV infusion of AMG 553
  Interventions: Drug: AMG 553

INTERVENTIONS:
Drug: AMG 553 — AMG 553 is a chimeric antigen T-cell receptor (CAR-T) therapy

SUMMARY:
Evaluate the safety and tolerability of AMG 553 in adult and adolescent subjects with FLT3-positive R/R AML.

Determine the maximum tolerated cell dose (MTCD) or recommended phase 2 cell dose (RP2CD) of AMG 553.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent/assent prior to initiation of any study-specific activities/procedures.
* Age greater than or equal to 12 years old at the time of signing the informed consent
* Relapsed/Refractory Acute Myeloid Leukemia (AML) as defined by the World Health Organization (WHO) Classification as persisting or recurring following 1 or more treatment courses (exceptions noted in exclusion criteria). Subjects must be intolerant to or ineligible for available therapies (eg, patients with FLT3 ITD/TKD mutations must have failed FLT3 inhibitors like midostaurin).
* FLT3 positivity: FLT3 expression on myeloblasts must be confirmed by local lab flow cytometry using an antibody targeting CD135 (FLT3)
* Myeloblasts greater than 5% in bone marrow and/or peripheral blood, as confirmed by immunophenotype by flow cytometry.
* Subject must have a donor or stem cell source identified for allogeneic transplantation, either related (7/8 or 8/8 allele matched or haploidentical), unrelated (7/8 or 8/8 allele matched donor), or cord blood stem cell source (at least 4/6 matched).
* Karnofsky performance score greater than or equal to 50 (for subjects aged greater than or equal to 16 years) or Lansky (for subjects aged less than 16 years) performance score greater than or equal to 50.
* Adequate organ function, defined as follows: Coagulation function: prothrombin timeprothrombin time/international normalization ratio (PT/INR) and partial thromboplastin time (PTT) less than or equal to 1.5 x Institutional Upper Limit of Normal Renal function as follows: Estimated Glomerular filtration rate by institutional formula greater than 60 mL/min/1.73 m2 or serum creatinine less than 2 times upper limit of normal (ULN) for the subject's age. Hepatic function: aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase less than 3 X upper limit of normal ULN. Total bilirubin less than 1.5 X upper limit of normal ULN. Cardiac function: Cardiac ejection fraction greater than or equal to 50%, no evidence of pericardial effusion as determined by an echocardiogram or Multigated Acquisition (MUGA) scan, and no clinically significant ECG findings.

Exclusion Criteria:

* Subjects with acute promyelocytic leukemia (APML).
* Active extramedullary AML in the central nervous system (CNS).
* Subjects with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the Amgen Medical Monitor.
* History of Down syndrome or any DNA fragility syndromes such as Bloom's syndrome.
* Autologous hematopoietic stem cell transplant (HSCT) within 6 weeks prior to enrollment
* Allogeneic hematopoietic stem cell transplant (HSCT) within 3 months prior to enrollment
* Any graft-versus-host disease requiring systemic therapy with immunomodulators
* Subjects with history or presence of clinically relevant non-malignant CNS disease requiring treatment (eg, uncontrolled seizures)
* Subjects with clinically relevant or uncontrolled active infections
* History or evidence of significant cardiovascular risk including any of the following: symptomatic congestive heart failure, unstable angina, clinically significant arrhythmias (eg, ventricular fibrillation, ventricular tachycardia etc.), coronary angioplasty within 6 months before dosing, intra-cardiac defibrillators or any clinically relevant concurrent disorder that may pose a risk to subject safety or interfere with study evaluation, procedures, or completion.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 3 months prior to enrollment.
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months before enrollment.
* Positive test for human immunodeficiency virus (HIV)
* Positive for hepatitis B surface antigen (HepBsAg)
* Positive for acute or chronic hepatitis C. Exceptions: Acute hepatitis C and completely cleared of the virus (demonstrated by negative viral load). Chronic hepatitis C with undetectable viral load defined by sustained virologic response 24 weeks (SVR24) after completion of anti-hepatitis C treatment.
* Received live vaccine(s) within 4 weeks of enrollment.
* Unresolved toxicities from prior antitumor therapy not having resolved to Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 grade 1 with the exception of myelosuppression (eg, neutropenia, anemia, thrombocytopenia) or are stable and well controlled AND there is agreement to allow by both the investigator and sponsor.
* Treatment with systemic immune modulators including, but not limited to, non-topical systemic corticosteroids, cyclosporine, and tacrolimus within 2 weeks before enrollment (exception: low dose systemic corticosteroids if used for blood transfusion reactions or similar).
* Major surgery within 28 days of enrollment with the exception of biopsy and insertion of central venous catheter.
* Subject has known sensitivity and immediate hypersensitivity to any components of AMG 553 or lymphodepleting regimen (cyclophosphamide and fludarabine).
* Other anti-cancer therapy (eg, investigational therapy, chemotherapy, antibody therapy, molecular targeted therapy) within 14 days (or 5 half-lives, whichever is shorter) prior to leukapheresis. Use of immune checkpoint inhibitors is excluded 3 months prior to leukapheresis.
* Prior treatment with any CAR-T or other genetically modified cell therapy.
* Presence of any clinically relevant indwelling line or drain (eg, percutaneous nephrostomy tube, biliary drain, or pleural/peritoneal/pericardial catheter).
* History of autoimmune disease (eg, Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years prior to enrollment.
* Females of child-bearing potential who are not willing to practice a highly effective method(s) of birth control from the time of consent through 6 months after AMG 553 infusion day.
* Females who are pregnant or planning to become pregnant or breastfeeding or who plan to breastfeed from the time of consent through 6 months after AMG 553 infusion day.
* Males who are unwilling to abstain from sperm donation while on study through 6 months after AMG 553 infusion day.
* Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception from the time of consent through 6 months after AMG 553 infusion day.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Subjects with clinically significant pre-existing liver disease, such as cirrhosis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-13 (Estimated); Primary Completion 2030-08-07 (Estimated); Study Completion 2030-08-07 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 3 Months
Treatment-emergent adverse events | 3 months
Treatment-related adverse events | 3 months

SECONDARY OUTCOMES:
Complete response (CR) | 3 months
  Evidence of anti-leukemic activity of AMG 553
Complete response with partial recovery of peripheral blood counts (CRh) | 3 months
  Evidence of anti-leukemic activity of AMG 553
Complete response with incomplete recovery of peripheral blood counts (CRi) | 3 months
  Evidence of anti-leukemic activity of AMG 553
Morphologic leukemia-free state (MLFS) | 3 months
  Evidence of anti-leukemic activity of AMG 553
Duration of response (DOR) | 3 months
  Evidence of anti-leukemic activity of AMG 553
Progression free survival (PFS) | 3 months
  Evidence of anti-leukemic activiy of AMG 553
Overall Survival (OS) | 3 months
  Evidence of anti-leukemic activity of AMG 553
Proportion of subjects with minimal-residual disease (MRD) negative response | 3 Months
  Evaluated proportion of subjects with minimal residual disease (MRD) negative response measured by flow cytometry in subjects achieving morphologic response defined by complete response (CR), complete response with partial recovery of peripheral blood counts (CRh), complete response with incomplete recovery of peripheral blood counts (CRi) measured by modified International Working Group (IWG) criteria.
The area under the concentration time-curve (AUC) of AMG 553 | 3 Months
  Evaluate the cellular kinetics of AMG 553 post infusion
Peak levels of AMG 553 (maximum concentration or Cmax) | 3 months
  Evaluate the cellular kinetics of AMG 553 post infusion

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Stanford University, Palo Alto, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com